CLINICAL TRIAL: NCT00508586
Title: A Phase 1b Study to Assess the Safety, Feasibility, Pharmacokinetics, and Activity of PTC299 Monotherapy or Combination Therapy With Hormonal Agents in Patients With Metastatic Breast Cancer
Brief Title: PTC299 and Hormonal Agent for Treatment of Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC299-ONC-003-BRC; BC050203
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; PTC299; VEGF; Angiogenesis; Post-transcriptional control; Aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — emvododstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PTC299 with an aromatase inhibitor
  Interventions: Drug: PTC299

INTERVENTIONS:
Drug: PTC299 — PTC299 orally administered twice per day given in combination with anastrozole (Arimidex®), letrazole (Femara®), or exemestane (Aromasin®)

SUMMARY:
Formation of new blood vessels (angiogenesis) is important for tumor growth in metastatic breast cancer. It is known that tumors make a protein called vascular endothelial growth factor (VEGF) and there are higher levels of VEGF in the tumors and blood of many women with metastatic breast cancer. VEGF stimulates the formation of blood vessels that supply the tumor with nutrients and oxygen. PTC299 is an oral drug that has been shown to decrease production of VEGF in animal models of human cancer. In these animal models, oral PTC299 administration decreases VEGF levels in the tumor and in the bloodstream, decreases blood vessel numbers in the tumor, and significantly slows or halts tumor growth. Safety studies in research animals indicate good tolerability at doses and drug levels that are higher than those planned for the clinical studies. Results from Phase 1a studies in healthy volunteers indicate that PTC299 achieves levels of PTC299 in the bloodstream that are known to be active in animal models of human cancer. This Phase 1b study is designed to test the hypothesis that PTC299 will be tolerable and will show evidence of VEGF reduction and antitumor activity when administered orally in combination with anastrozole (Arimidex®), letrozole (Femara®), or exemestane (Aromasin®) to women with metastatic breast cancer.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages. In Stage 1 of the study, successive groups of 3 to 6 patients will receive progressively higher PTC299 dose levels; in this stage, treatment will be given in repeated 6-week cycles consisting of 4 weeks of oral PTC299 twice per day followed by a 2-week, no-drug period. During Stage 2, study candidates must be women with natural or induced suppression of ovarian function to post-menopausal levels who are receiving or are candidates for hormonal therapy. These subjects will receive continuous administration of PTC299, 100 mg/dose BID, in repeated 6-week cycles in combination with continuous administration of one of 3 hormonal agents. All planned PTC299 dose levels in all stages are expected to achieve circulating blood levels of PTC299 known to be active in animal models of human cancer. Treatment for each patient can continue as long as the therapy appears to be safely offering tumor control to that patient. Up to 36 evaluable patients will be accrued across both stages.

ELIGIBILITY:
Major Eligibility Criteria:

1. Female sex.
2. Age ≥18 years.
3. Body weight 40-100 kg.
4. ECOG performance status of 0 or 1.
5. Histologically or cytologically confirmed adenocarcinoma of the breast.
6. Presence of metastatic disease not amenable to surgery, radiation therapy, or chemoradiotherapy with curative intent.
7. No active second metastatic malignancy other than breast cancer.
8. No unstable brain or leptomeningeal disease.
9. Discontinuation of other therapies (except for anastrozole, letrozole, or exemestane) for the treatment of breast cancer and resolution of any acute toxic effects of prior therapies.
10. Adequate bone marrow, liver, and kidney function.
11. No uncontrolled hypertension, major bleeding, HIV infection or recent acute cardiovascular event.
12. If sexually active and not postmenopausal or surgically sterile, willingness to abstain from sexual intercourse or employ an effective barrier method of contraception during the study drug administration and follow-up periods.
13. No pregnancy or breast-feeding.
14. Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
15. Willingness to provide informed consent. In addition to the criteria noted above, Stage 2 subjects must also have natural or induced suppression of ovarian function to post-menopausal levels and be receiving or be a candidate for hormonal therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) within the tested dose range. | 6 Weeks

SECONDARY OUTCOMES:
Overall safety profile | 6 Weeks
Study drug compliance | 6 Weeks
Pharmacokinetics | 6 Weeks
Circulating angiogenic markers | 6 Weeks
Tumor perfusion as assessed by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) | 6 Weeks
Tumor metabolism as assessed by fluorodeoxyglucose positron emission tomography (FDG-PET) | 6 Weeks
Antitumor activity as assessed by computed tomography (CT) scans and tumor markers | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Barth, MD, Study Director — PTC Therapeutics, Inc.
Locations (3):
- United States (3):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - New York University Clinical Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: PTC Therapeutics, Inc. web site — http://www.ptcbio.com